CLINICAL TRIAL: NCT01738698
Title: A Phase 3 Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, 12-week, Forced-dose Titration Study to Evaluate the Efficacy, Safety, and Tolerability of SPD489 40mg, 100mg, or 160mg as Adjunctive Treatment to Established Maintenance Doses of Antipsychotic Medications on Negative Symptoms in Clinically Stable Adults Who Have Persistent Predominant Negative Symptoms of Schizophrenia
Brief Title: Adjunctive SPD489 to Antipsychotic Medication in Clinically Stable Adults With Persistent Predominant Negative Symptoms of Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-338; 2012-003918-14 (EudraCT Number)
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SPD489 40mg (Experimental)
  Interventions: Drug: SPD489 40mg
- SPD489 100mg (Experimental)
  Interventions: Drug: SPD489 100mg
- SPD489 160mg (Experimental)
  Interventions: Drug: SPD489 160mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD489 40mg — Oral administration of 40 mg once-daily for up to 12 weeks
  Other Names: lisdexamfetamine dimesylate, LDX, Vyvanse
  Arms: SPD489 40mg
Drug: SPD489 100mg — Oral administration of 100 mg once-daily for up to 12 weeks
  Other Names: lisdexamfetamine dimesylate, LDX, Vyvanse
  Arms: SPD489 100mg
Drug: SPD489 160mg — Oral administration of 160 mg once-daily for up to 12 weeks
  Other Names: lisdexamfetamine dimesylate, LDX, Vyvanse
  Arms: SPD489 160mg
Drug: Placebo — Oral administration once-daily for 12 weeks
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine whether SPD489 40 mg, 100 mg, and 160 mg are effective and safe in the treatment of Negative Symptoms of Schizophrenia (NSS).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Has a reliable informant (eg, family member, social worker, caseworker, or nurse that spends >4 hours/week with the subject)
* Fixed home/place of residence and can be reached by telephone
* On a stable dose of antipsychotic medications
* Able to swallow capsules

Exclusion Criteria:

* Taking lithium, carbamazepine, lamotrigine, gabapentin, cholinesterase inhibitors, modafinil, or other stimulants such as methylphenidate and other amphetamine products
* Treated with clozapine in past 30 days
* Lifetime history of stimulant, cocaine, or amphetamine abuse or dependence
* History of seizures (other than infantile febrile seizures), any tic disorder, or current diagnosis and/or a known family history of Tourette's Disorder, serious neurological disease, history of significant head trauma, dementia, cerebrovascular disease, Parkinson's disease, or intracranial lesions
* Uncontrolled hypertension
* History of thyroid disorder that has not been stabilized on thyroid medication
* Glaucoma
* Pregnant or nursing
* Subject has received an investigational product or participated in a clinical study within 30 day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2013-04-01 (Actual); Study Completion 2013-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- University Hills Clinical Research, Irving, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Period: Overall Study
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Negative Symptom Assessment - 16-item (NSA-16) Total Score at 12 Weeks
Time Frame: Baseline and 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in the Personal and Social Performance Scale (PSP) Score at 12 Weeks
Time Frame: Baseline and 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score at 12 Weeks
Time Frame: Baseline and 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Barnes Akathisia Scale (BAS) Total Score at 12 Weeks
Time Frame: Baseline and 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Amphetamine Cessation Symptom Assessment (ACSA) Total Score at 12 Weeks
Time Frame: Baseline and 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in the Abnormal Involuntary Movement Scale (AIMS) at 12 Weeks
Time Frame: Baseline and 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Scores at 12 Weeks
Time Frame: Baseline and 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at 12 Weeks
Time Frame: Baseline and 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Social Functioning Scale (SFS) at 12 Weeks
Time Frame: Baseline and 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline in Clinical Evaluation of Harmful Behavior (CEHB) Scale at 12 Weeks
Time Frame: Baseline and 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Clinical Global Impression-Schizophrenia Severity of Illness (CGI-SCH-S) Scale
Time Frame: Baseline and week 12
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Clinical Global Impression-Schizophrenia Degree of Change (CGI-SCH-C) Scale
Time Frame: Up to 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Time Frame: Up to 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline in Calgary Depression Scale for Schizophrenia (CDSS) at 12 Weeks
Time Frame: Baseline and 12 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Ambulatory Blood Pressure Monitoring (ABPM)
Time Frame: Baseline and Weeks 4 and 10
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 40mg | SPD489 100mg | SPD489 160mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.